CLINICAL TRIAL: NCT02620527
Title: Study of Concordance Between Circulating Tumor DNA Assay and Foundation One Tissue Analysis For Genomic Alterations
Brief Title: Concordance Between ctDNA Assay and FoundationOne
Status: Completed | Type: Observational
Sponsor: Foundation Medicine (Industry)
Collaborators: Johns Hopkins University (Other); Oncology Consultants (Unknown); Comprehensive Blood and Cancer Center (Other); Illinois CancerCare (Other); Sanford Health (Other); Eastchester Center for Cancer Care (Other); Rutgers Cancer Institute of New Jersey (Other); Cone Health (Other); Nebraska Cancer Specialists (Unknown); University of California, Davis (Other); University of Chicago (Other); Northeast Georgia Medical Center (Unknown); Hematology Oncology Associates of Fredericksburg (Unknown); Memorial Sloan Kettering Cancer Center (Other); Oncology Hematology Care, Inc (Unknown); Montefiore Medical Center (Other); Quincy Medical Group (Other); Prisma Health-Upstate (Other); Mary Crowley Cancer Research Center (Unknown); Texas Health (Unknown); University of California, San Diego (Other); Avera Cancer Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: FMI-CTDNA-15
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Circulating Tumor DNA; Cancer; Neoplasms; Genomic Testing; Genomic Alterations
Keywords: Circulating Tumor DNA; Cancer; Neoplasms; Genomic Testing; FoundationOne; Cell Free DNA; ctDNA; cfDNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Foundation Medicine Inc. (FMI) is interested in studying the concordance of genomic alterations between primary and/or metastatic surgical biopsies, and circulating tumor DNA (ctDNA) within different solid tumor types and has been developing an assay in order to do so.

DETAILED DESCRIPTION:
The purpose of this study is to assess whether a new ctDNA assay developed by Foundation Medicine is able to detect genomic alterations in peripheral blood that are consistent with the genomic alterations detected in a patient's matched primary and/or metastatic tumor biopsy sample analyzed by the FoundationOne® test. Study sites will provide matched solid tumor and peripheral blood samples of cancer patients to FMI for the purpose of testing the concordance of the FMI ctDNA assay to the FoundationOne® test. Participation in this study is part of a broader 2000 patient study to determine which tumor types are most readily measured via ctDNA profiling, and to learn of the similarity between the alterations found in a patient's tumor biopsy and the ctDNA from their blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a solid tumor biopsy isolated for analysis by FoundationOne under their standard clinical care

Exclusion Criteria:

* Tumor specimens where no cancer representative of the diagnosis is found in submitted tissue
* Tumor specimens where insufficient DNA (<50 ng) is provided to run the FoundationOne test.
* Tumor specimens with ≤20% tumor nuclei (all specimens).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cancer and who have had a solid tumor biopsy isolated for analysis by FoundationOne
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Whether new ctDNA assay can detect genomic alterations in peripheral blood that are consistent with those detected by FoundationOne in matched solid tumor samples | 6-12 months
Determine which tumor types are most amenable to detection using peripheral blood ctDNA assay | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Phil Stephens, PhD, Principal Investigator — Foundation Medicine
Locations (1):
- Foundation Medicine, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Zhou C, Yuan Z, Ma W, Qi L, Mahavongtrakul A, Li Y, Li H, Gong J, Fan RR, Li J, Molmen M, Clark TA, Pavlick D, Frampton GM, Forcier B, Moore EH, Shelton DK, Cooke M, Ali SM, Miller VA, Gregg JP, Stephens PJ, Li T. Clinical utility of tumor genomic profiling in patients with high plasma circulating tumor DNA burden or metabolically active tumors. J Hematol Oncol. 2018 Nov 6;11(1):129. doi: 10.1186/s13045-018-0671-8. PMID 30400986